CLINICAL TRIAL: NCT04974151
Title: Comparative Efficacy of Amlodipine Folic Acid vs. Amlodipine on the Risk of First Ischemic Stroke Among Participants With Hypertension and MTHFR 677 TT Genotype: A Multi-center, Randomized, Double-blind, Triple-dummy, Controlled Clinical Trial
Brief Title: China Stroke Primary Prevention Trial 2 for Participants With Hypertension and MTHFR 677 TT Genotype
Acronym: CSPPT2-TT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shenzhen Ausa Pharmed Co.,Ltd (Industry)
Collaborators: Peking University First Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); The First People's Hospital of Lianyungang (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Lianyungang Oriental Hospital (Other); Tengzhou Central People's Hospital (Other Government); The First Affiliated Hospital of Bengbu Medical University (Other); Shenzhen Prospective Medical Technology Co., LTD (Unknown); Weinan Central Hospital (Other); The First Affiliated Hospital of HuNan University of Medicine (Unknown); Loudi Central Hospital (Other); Yancheng First People's Hospital (Other); TAIHE country people's hospital (Unknown); First Affiliated Hospital of Gannan Medical University (Other); Yangjiang People's Hospital (Other); Deyang People's Hospital (Other); Bozhou people's hospital (Unknown); Chizhou people's hospital (Unknown); Lianyungang Second People's Hospital (Unknown); The Affiliated Hospital Of Southwest Medical University (Other); Chengdu Fifth People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPPT2-TT_2020
Record Dates: First submitted 2021-07-13; First posted 2021-07-23 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Hypertension; MTHFR 677 TT Genotype
Keywords: Folic acid; Homocysteine; MTHFR 677 TT genotype; Randomized controlled trial; Ischemic stroke; 5-MTHF
MeSH Terms: conditions — Hypertension; Ischemic Stroke | interventions — Amlodipine; Folic Acid; 5-methyltetrahydrofolate

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, controlled, double-blind, triple-dummy clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Amlodipine (5mg/d) (Active Comparator): Amlodipine 5mg x1 tablet + Amlodipine folic acid (dummy) x1 tablet + 5-MTHF (dummy) x2 tablets, taken orally, in the morning after waking up.
  Amlodipine tablets, amlodipine folic acid placebos, and 5-MTHF placebos are provided in aluminum-plastic blister plate. Each package includes 100 days of treatment drug (including 10 extra days of treatment for the follow-up window). A package of medication consists of 50 plates, each plate includes a total of 8 tablets arranged as follows: amlodipine 5mg x2 tablets + amlodipine folic acid (dummy) x2 tablets + 5-MTHF (dummy) x4 tablets. Affixed to the package is the randomized treatment drug label (400 tablets/package, 4 tablets/day).
  Interventions: Drug: Amlodipine besylate; Drug: Amlodipine folic acid placebo; Drug: 5-MTHF Placebos
- Amlodipine folic acid (5.8mg/d) (Experimental): Amlodipine folic acid 5.8mg x1 tablet + amlodipine (dummy) x1 tablet + 5-MTHF (dummy) x2 tablets, taken orally, in the morning after waking up.
  Amlodipine folic acid tablets, amlodipine placebos, and 5-MTHF placebos are provided in aluminum-plastic blister plate. Each package includes 100 days of treatment drug (including 10 extra days of treatment for the follow-up window). A package of medication consists of 50 plates, each plate includes a total of 8 tablets arranged as follows: amlodipine folic acid 5.8mg x2 tablets + amlodipine (dummy) x2 tablets + 5-MTHF (dummy) x4 tablets. Affixed to the package is the randomized treatment drug label (400 tablets/package, 4 tablets/day).
  Interventions: Drug: Amlodipine besylate And Folic Acid; Drug: Amlodipine placebo; Drug: 5-MTHF Placebos
- Amlodipine folic acid (5.8mg/d) + 5-MTHF (0.4mg/d) (Experimental): Amlodipine folic acid 5.8mg x1 tablet + 5-methyltetrahydrofolate 0.2mg x2 tablets + amlodipine (dummy) x1 tablet, taken orally, in the morning after waking up.
  Amlodipine folic acid tablets, 5-MTHF, and amlodipine placebos are provided in aluminum-plastic blister plate. Each package includes 100 days of treatment drug (including 10 extra days of treatment for the follow-up window). A package of medication consists of 50 plates, each plate includes a total of 8 tablets arranged as follows: amlodipine folic acid 5.8mg x2 tablets + amlodipine (dummy) x2 tablets + 5-MTHF, 0.2mg x4 tablets. Affixed to the package is the randomized treatment drug label (400 tablets/package, 4 tablets/day).
  Interventions: Drug: Amlodipine besylate And Folic Acid; Drug: 5-methyltetrahydrofolate (5-MTHF); Drug: Amlodipine placebo

INTERVENTIONS:
Drug: Amlodipine besylate — The amlodipine used in this study is a listed product.
  Other Names: Amlodipine
  Arms: Amlodipine (5mg/d)
Drug: Amlodipine besylate And Folic Acid — The amlodipine besylate and folic acid tablets have been approved for listing by the China Food and Drug Administration, approval number: Zhunzi H20180020.
  Other Names: Amlodipine Folic Acid; Anye
  Arms: Amlodipine folic acid (5.8mg/d); Amlodipine folic acid (5.8mg/d) + 5-MTHF (0.4mg/d)
Drug: 5-methyltetrahydrofolate (5-MTHF) — The 5-MTHF used in this study is a listed product.
  Other Names: 5-MTHF
  Arms: Amlodipine folic acid (5.8mg/d) + 5-MTHF (0.4mg/d)
Drug: Amlodipine placebo — Amlodipine placebos are dummy pills of amlodipine with identical appearance.
  Other Names: Amlodipine (dummy)
  Arms: Amlodipine folic acid (5.8mg/d); Amlodipine folic acid (5.8mg/d) + 5-MTHF (0.4mg/d)
Drug: Amlodipine folic acid placebo — Amlodipine folic acid placebos are dummy pills of amlodipine folic acid with identical appearance.
  Other Names: Amlodipine folic acid (dummy)
  Arms: Amlodipine (5mg/d)
Drug: 5-MTHF Placebos — 5-MTHF placebos are the dummy pills of 5-MTHF with identical appearance.
  Other Names: 5-MTHF (dummy)
  Arms: Amlodipine (5mg/d); Amlodipine folic acid (5.8mg/d)

SUMMARY:
This is a multi-center, randomized, double-blind, triple-dummy, controlled trial in 24,000 Chinese men and women with hypertension and MTHFR 677 TT genotype.

The study participants will be randomized to one of the three treatment groups:

Group A: amlodipine tablet (5mg), taken orally, once daily, serving as active comparator.

Group B: amlodipine folic acid 5.8mg tablet (5mg amlodipine and 0.8mg folic acid), taken orally, once daily.

Group C: amlodipine folic acid 5.8mg tablet plus 5-methyltetrahydrofolate (5-MTHF, 0.4mg), taken orally, once daily.

The primary endpoint is first ischemic stroke.

DETAILED DESCRIPTION:
This study consists of 3 periods: Screening, Run-in, and Randomized treatment.

Period I: Screening (V0)

The purpose of Period I is to obtain informed consent and screen for eligible participants.

After obtaining written informed consent, at the screening visit (V0), participants will complete a face-to-face interview and clinical evaluation and measurements. Their biological samples will be collected for laboratory analyses. Collectively, these information will help to determine eligibility for inclusion in the study.

Period II: Run-in Period (VD)

The purpose of Run-in is to assess participants' compliance for following the amlodipine treatment regimen as well as to observe participants' tolerance to amlodipine, so as to screen out those with poor compliance or intolerance to amlodipine treatment.

The run-in phase lasted 2 to 4 weeks, during which oral administration of Amlodipine tablets (5 mg) was given once daily.

Period III: Randomized Treatment (V1-V21)

This is a 5-year period of randomized, double-blind, triple-dummy, controlled treatment. At each of the research centers, participants who remain eligible for participation in the study will be randomized into 3 treatment groups:

A. Amlodipine-only (5mg/d) with an amlodipine folic acid placebo and 5-MTHF placebos.

B. Amlodipine folic acid tablet (5.8mg/d) with amlodipine placebo and 5-MTHF placebo.

C. Amlodipine folic acid tablets (5.8mg/d) and 5-MTHF (0.4mg/d) with an amlodipine placebo in a 1:1:1 ratio, using the randomization and trial supply management (RTSM) platform.

During the treatment period, other antihypertensive drugs can be added to achieve blood pressure control (BP ≤140/90mmHg), including Valsartan (80mg/d), or/and Indapamide (1.5mg/d), or/and metoprolol tartrate tablets (25mg/d). Participants will be followed up every 3 months during the treatment period, and the treatment drugs will be distributed at each visit.

A total of 24,000 participants will be randomly assigned to one of three treatment groups (Group A n=8,000, Group B n=8,000, Group C n=8,000). Based on published data from CSPPT (Huo et al, JAMA, 2015), the 5-year cumulative incidence of first ischemic stroke in the amlodipine-only group is 3.5%. Assuming the 5-year cumulative incidence of first ischemic stroke in the amlodipine-only group is around 3.5%, this trial has 80% power to detect a 20% difference between group A and group B+C in the observed hazard ratio (HR) for incident ischemic stroke (HR≤0.80), at a two-sided significance level of α=0.05. If instead, the 5-year incidence of ischemic stroke in the amlodipine-only group is 2.5%, this trial has 80% power to detect a 23% difference between the treatment groups (A vs B+C) (HR≤0.77).

There are two planned interim analyses, one at the end of the third year, and another at the end of the fourth year. The O'Brien-Fleming alpha-spending function will be used to define the significance level of each interim analysis to ensure that the final overall two-sided significance level of α=0.05 is met.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged ≥45 and <75 years.
2. Hypertension: Previously diagnosed with primary hypertension and has been taking antihypertensive medication within the past two weeks; OR has not been taking antihypertensive medications within the last two weeks, but meets the following criteria for hypertension: SBP≥140 mmHg and/or DBP≥90 mmHg (average of at least 2 measurements each time) at two separate (not on the same day) clinical visits.
3. MTHFR 677 TT genotype (based on the test results from the central laboratory during the screening period or a previous official test report from a laboratory with medical testing qualifications).
4. Voluntarily participates and has given signed informed consent.

Randomized-treatment phase inclusion criteria:

1. Good compliance during the run-in period, and unlikely to discontinue treatment;
2. No stroke or cardiovascular events during the run-in period;
3. The participant voluntarily agrees to continue the study.

Exclusion Criteria:

1. Previously diagnosed secondary hypertension;
2. Previously diagnosed stroke;
3. Previously diagnosed myocardial infarction;
4. Previously diagnosed heart failure;
5. Previously diagnosed atrial fibrillation;
6. Cardio-cerebral-kidney revascularization and/or other large arterial stent;
7. Currently on dialysis, or diagnosed with stage 4-5 chronic kidney disease, or eGFR <30 mL/ min/1.73m²;
8. Known to have congenital (such as aortic stenosis) or acquired organic heart disease;
9. Known to have any of the following severe diseases or conditions:

   1. Digestive system: i. Previously diagnosed with any form of viral hepatitis that is currently still in the active phase; ii. Abnormal liver function test before enrollment (any of ALT, AST, GGT, TBIL, DBIL test 3 times higher than normal, or ALB≤30g/L); iii. Subtotal gastrectomy and/or gastrojejunostomy;
   2. Respiratory system: previously diagnosed with pulmonary heart disease;
   3. Presence of malignant tumors or other severe diseases;
   4. Presence of long-term gastrointestinal symptoms such as ; anorexia, decreased appetite, nausea, and abdominal bloating;
   5. Previously diagnosed with vitamin B12 deficiency and/or its related diseases.
10. Participant, at the investigator's discretion, is assessed to be unsuitable for the study, for reasons including but not limited to the presence of abnormal laboratory results, or clinical conditions;
11. Prior history of significant intolerance due to adverse reactions resulting from usage of amlodipine or other CCBs, valsartan or other ARBs, indapamide or other similar diuretics, metoprolol tartaric acid or other beta-blockers, or any drugs or health products containing folate or folic acid;
12. Regular consumption of folic acid or vitamin B compounds, or other compounds containing folic acid in the past 3 months;
13. The presence of any of the following conditions that could negatively influence a participant's ability to consent or participate in the trial:

    1. Dementia;
    2. Severe mental disorders;
    3. Inability to express informed consent;
    4. Unlikely to complete the study follow-up as specified by the protocol, or plans to relocate outside of the study area in the near future;
    5. History of poor compliance when taking antihypertensive medications or is expected to have poor compliance during the study;
14. Refusal to participate, or inability to modify current drug regimen;
15. Women who are pregnant or breastfeeding; or subjects of childbearing potential who are unwilling or unable to use effective contraception during the study period.
16. Within one month prior to the first visit, having participated in any clinical trial for a drug that has not yet been officially approved by the state or is not currently approved for sale; or currently participating in any clinical trial that could potentially impact the results of this study (medication use, drug efficacy, drug interaction, etc.).

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24000 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
First ischemic stroke | By the end of the fifth year of the study
  The primary aim of the trial is to determine whether amlodipine folic acid tablets (including Group B and Group C), compared to amlodipine alone (Group A), can further reduce the risk of first ischemic stroke among eligible participants with hypertension and the MTHFR 677 TT genotype.

SECONDARY OUTCOMES:
First ischemic stroke (for refined treatment group comparisons) | By the end of the fifth year of the study
  We will examine whether there exist significant differences in efficacy in reducing the risk of first ischemic stroke between the following pairs of treatment groups:
  Group B vs. Group A
  Group C vs. Group A
  Group B vs. Group C
First stroke (ischemic and hemorrhagic) | By the end of the fifth year from baseline
  We will examine whether there exist significant differences in efficacy in reducing the risk of first stroke between the following pairs of treatment groups:
  Groups B + C vs. Group A
  Group B vs. Group A
  Group C vs. Group A
  Group B vs. Group C
Composite cardiovascular endpoint (first non-fatal stroke, first non-fatal myocardial infarction, cardiovascular death) | By the end of the fifth year from baseline
  We will examine whether there exist significant differences in efficacy in reducing the risk of composite cardiovascular endpoint between the following pairs of treatment groups:
  Groups B + C vs. Group A
  Group B vs. Group A
  Group C vs. Group A
  Group B vs. Group C
Kidney outcomes | By the end of the fifth year from baseline
  1. The primary kidney outcome is composite kidney outcome, defined as: (1) a decrease in eGFR of 30% or more and to a level of less than 60 mL/min/1.73 m2 if the baseline eGFR is 60 mL/min/1.73 m2 or more, or (2) a decrease in eGFR of 50% or more if the baseline eGFR is less than 60 mL/min/1.73 m2, or (3) end-stage kidney disease (ESKD) (eGFR <15 mL/min/1.73m2 or dialysis or kidney transplantation).
  2. Secondary kidney outcomes: (1) eGFR decline ≥40% from baseline, or end-stage kidney disease; (2) annual rate of relative decline in eGFR; (3) Incidence of proteinuria, or progression of proteinuria.
  We will examine whether there exist significant differences in treatment efficacy on the above kidney endpoints between the following pairs of treatment groups:
  Groups B + C vs. Group A
  Group B vs. Group A
  Group C vs. Group A
  Group B vs. Group C
First hemorrhagic stroke | By the end of the fifth year from baseline
  We will examine whether amlodipine folic acid tablets (including Groups B and C), compared to amlodipine alone (Group A), show significantly greater efficacy in preventing first hemorrhagic stroke.
First myocardial infarction | By the end of the fifth year from baseline
  We will examine whether amlodipine folic acid tablets (including Groups B and C), compared to amlodipine alone (Group A), show significantly greater efficacy in preventing first myocardial infarction.
First coronary revascularization (coronary artery bypass grafting [CABG] or percutaneous coronary intervention [PCI]) | By the end of the fifth year from baseline
  We will examine whether amlodipine folic acid tablets (including Groups B and C), compared to amlodipine alone (Group A), show significantly greater efficacy in preventing first coronary revascularization.
Cardiovascular death | By the end of the fifth year from baseline
  We will examine whether amlodipine folic acid tablets (including Groups B and C), compared to amlodipine alone (Group A), show significantly greater efficacy in preventing cardiovascular death.

OTHER OUTCOMES:
Malignant tumors | By the end of the fifth year of the study
  We will examine whether there exist significant differences in efficacy in reducing the risk of malignant tumors between the Groups B + C and Group A.
All-cause mortality | By the end of the fifth year of the study
  We will examine whether there exist significant differences in efficacy in reducing the risk of all-cause mortality between the Groups B + C and Group A.
Blood pressure levels | 1) Blood pressure levels at one year, three-year and at the end of follow-up(up to 5 years). 2) Average blood pressure levels across all visits in the first and third years of follow-up, as well as for the entire follow-up period (up to 5 years).
  We will examine whether there exist significant differences in treatment efficacy on the blood pressure levels between the following pairs of treatment groups:
  Groups B + C vs. Group A
  Group B vs. Group A
  Group C vs. Group A
  Group B vs. Group C
Blood pressure variability | 1) Average blood pressure variability across all visits in the first and third years of follow-up, and across all visits throughout the entire follow-up period (up to 5 years).
  We will examine whether there exist significant differences in treatment efficacy on the blood pressure variability between the following pairs of treatment groups:
  Groups B + C vs. Group A
  Group B vs. Group A
  Group C vs. Group A
  Group B vs. Group C
Blood pressure target achievement rates | 1) Blood pressure target achievementrates at 1-year, 3-year and at the end of follow-up(up to 5 years). 2) Average bloodpressure target achievement rates across all visits in the first and third years of follow-up, and for the entire follow-up period.]
  We will examine whether there exist significant differences in treatment efficacy on the blood pressure target achievement rates between the following pairs of treatment groups:
  Groups B + C vs. Group A
  Group B vs. Group A
  Group C vs. Group A
  Group B vs. Group C
Serum folate level | Serum folate levels at one year, three-year and at the end of follow-up(up to 5 years).
  We will examine whether there exist significant differences in treatment efficacy on the serum folate levels between the following pairs of treatment groups:
  Groups B + C vs. Group A
  Group B vs. Group A
  Group C vs. Group A
  Group B vs. Group C
Serum folate change | Serum folate changes at one year, three-year and at the end of follow-up(up to 5 years).
  We will examine whether there exist significant differences in treatment efficacy on the serum folate changes between the following pairs of treatment groups:
  Groups B + C vs. Group A
  Group B vs. Group A
  Group C vs. Group A
  Group B vs. Group C
Plasma tHcy level | Plasma total homocysteine levels at one year, three-year and at the end of follow-up(up to 5 years).
  We will examine whether there exist significant differences in treatment efficacy on the plasma total homocysteine levels between the following pairs of treatment groups:
  Groups B + C vs. Group A
  Group B vs. Group A
  Group C vs. Group A
  Group B vs. Group C
Plasma tHcy change | Plasma total homocysteine changes at one year, three-year and at the end of follow-up(up to 5 years).
  We will examine whether there exist significant differences in treatment efficacy on the plasma total homocysteine changes between the following pairs of treatment groups:
  Groups B + C vs. Group A
  Group B vs. Group A
  Group C vs. Group A
  Group B vs. Group C

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Li, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (20):
- China (20):
  - First Affillated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Bozhou People's Hospital, Bozhou, Anhui
  - Chizhou People's Hospital, Chizhou, Anhui
  - Taihe County People's Hospital, Fuyang, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Yangjiang People's Hospital, Yangjiang, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The First Affiliated Hospital of Hunan University of Medicine, Huaihua, Hunan
  - Loudi Central Hospital, Loudi, Hunan
  - Lianyungang Oriental Hospital, Lianyungang, Jiangsu
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - The Second People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Yancheng First People's Hospital, Yancheng, Jiangsu
  - The First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Weinan Central Hospital, Weinan, Shaanxi
  - Tengzhou Central People's Hospital, Zaozhuang, Shandong
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Deyang People's Hospital, Deyang, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kjeldsen SE, Julius S, Hedner T, Hansson L. Stroke is more common than myocardial infarction in hypertension: analysis based on 11 major randomized intervention trials. Blood Press. 2001;10(4):190-2. doi: 10.1080/08037050152669684. No abstract available. PMID 11800055
- [Background] Collaboration HLT. Lowering blood homocysteine with folic acid based supplements: meta-analysis of randomised trials. Homocysteine Lowering Trialists' Collaboration. BMJ. 1998 Mar 21;316(7135):894-8. PMID 9569395
- [Background] Homocysteine Lowering Trialists' Collaboration. Dose-dependent effects of folic acid on blood concentrations of homocysteine: a meta-analysis of the randomized trials. Am J Clin Nutr. 2005 Oct;82(4):806-12. doi: 10.1093/ajcn/82.4.806. PMID 16210710
- [Background] Wilcken B, Bamforth F, Li Z, Zhu H, Ritvanen A, Renlund M, Stoll C, Alembik Y, Dott B, Czeizel AE, Gelman-Kohan Z, Scarano G, Bianca S, Ettore G, Tenconi R, Bellato S, Scala I, Mutchinick OM, Lopez MA, de Walle H, Hofstra R, Joutchenko L, Kavteladze L, Bermejo E, Martinez-Frias ML, Gallagher M, Erickson JD, Vollset SE, Mastroiacovo P, Andria G, Botto LD. Geographical and ethnic variation of the 677C>T allele of 5,10 methylenetetrahydrofolate reductase (MTHFR): findings from over 7000 newborns from 16 areas world wide. J Med Genet. 2003 Aug;40(8):619-25. doi: 10.1136/jmg.40.8.619. No abstract available. PMID 12920077
- [Background] Qin X, Li J, Cui Y, Liu Z, Zhao Z, Ge J, Guan D, Hu J, Wang Y, Zhang F, Xu X, Wang X, Xu X, Huo Y. MTHFR C677T and MTR A2756G polymorphisms and the homocysteine lowering efficacy of different doses of folic acid in hypertensive Chinese adults. Nutr J. 2012 Jan 10;11:2. doi: 10.1186/1475-2891-11-2. PMID 22230384
- [Background] Qin X, Li J, Cui Y, Liu Z, Zhao Z, Ge J, Guan D, Hu J, Wang Y, Zhang F, Xu X, Wang X, Xu X, Huo Y. Effect of folic acid intervention on the change of serum folate level in hypertensive Chinese adults: do methylenetetrahydrofolate reductase and methionine synthase gene polymorphisms affect therapeutic responses? Pharmacogenet Genomics. 2012 Jun;22(6):421-8. doi: 10.1097/FPC.0b013e32834ac5e8. PMID 21869730
- [Background] Xu X, Li J, Sheng W, Liu L. Meta-analysis of genetic studies from journals published in China of ischemic stroke in the Han Chinese population. Cerebrovasc Dis. 2008;26(1):48-62. doi: 10.1159/000135653. Epub 2008 May 30. PMID 18511872
- [Background] Qin X, Li J, Zhang Y, Ma W, Fan F, Wang B, Xing H, Tang G, Wang X, Xu X, Xu X, Huo Y. Prevalence and associated factors of diabetes and impaired fasting glucose in Chinese hypertensive adults aged 45 to 75 years. PLoS One. 2012;7(8):e42538. doi: 10.1371/journal.pone.0042538. Epub 2012 Aug 3. PMID 22880024
- [Background] Dong Q, Tang G, He M, Cai Y, Cai Y, Xing H, Sun L, Li J, Zhang Y, Fan F, Wang B, Sun N, Liu L, Xu X, Hou F, Shen H, Xu X, Huo Y. Methylenetetrahydrofolate reductase C677T polymorphism is associated with estimated glomerular filtration rate in hypertensive Chinese males. BMC Med Genet. 2012 Aug 16;13:74. doi: 10.1186/1471-2350-13-74. PMID 22897803
- [Background] Huo Y, Li J, Qin X, Huang Y, Wang X, Gottesman RF, Tang G, Wang B, Chen D, He M, Fu J, Cai Y, Shi X, Zhang Y, Cui Y, Sun N, Li X, Cheng X, Wang J, Yang X, Yang T, Xiao C, Zhao G, Dong Q, Zhu D, Wang X, Ge J, Zhao L, Hu D, Liu L, Hou FF; CSPPT Investigators. Efficacy of folic acid therapy in primary prevention of stroke among adults with hypertension in China: the CSPPT randomized clinical trial. JAMA. 2015 Apr 7;313(13):1325-35. doi: 10.1001/jama.2015.2274. PMID 25771069
- [Background] Huang X, Li Y, Li P, Li J, Bao H, Zhang Y, Wang B, Sun N, Wang J, He M, Yin D, Tang G, Chen Y, Cui Y, Huang Y, Hou FF, Qin X, Huo Y, Cheng X. Association between percent decline in serum total homocysteine and risk of first stroke. Neurology. 2017 Nov 14;89(20):2101-2107. doi: 10.1212/WNL.0000000000004648. Epub 2017 Oct 13. PMID 29030456
- [Background] Qin X, Li Y, Sun N, Wang H, Zhang Y, Wang J, Li J, Xu X, Liang M, Nie J, Wang B, Cheng X, Li N, Sun Y, Zhao L, Wang X, Hou FF, Huo Y. Elevated Homocysteine Concentrations Decrease the Antihypertensive Effect of Angiotensin-Converting Enzyme Inhibitors in Hypertensive Patients. Arterioscler Thromb Vasc Biol. 2017 Jan;37(1):166-172. doi: 10.1161/ATVBAHA.116.308515. Epub 2016 Nov 10. PMID 27834686